CLINICAL TRIAL: NCT06305130
Title: Prognostic Value of Eastern Cooperative Oncology Group Performance Status and American Society of Anesthesiologists Score in Patients Undergoing Radical Nephroureterectomy for Upper Tract Urothelial Carcinoma
Brief Title: Prognostic Value of Performance Scores in Patients Undergoing Surgery for Upper Tract Urothelial Carcinoma
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Hsin-Chih Yeh, Principal investigator, Kaohsiung Medical University
Other Study IDs: KMUHIRB-E(I)-20180214
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Carcinoma, Transitional Cell (RENI)
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary cohort (only one in this study): Patient data were collected from sixteen institutions across Taiwan, encompassing 6005 patients diagnosed with UTUC between 1988 and 2023. The study included all patients who underwent RNU with curative intent. After excluding those with incomplete data, a total of 2515 eligible patients were included in the final analysis.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Aim: to comprehensively evaluate the prognostic value of preoperative ECOG-PS scores and ASA scores in patients undergoing radical nephroureterectomy (RNU) for upper tract urothelial carcinoma.

Methods: multicentered cohort study

DETAILED DESCRIPTION:
Background:

The Eastern Cooperative Oncology Group (ECOG) performance status (PS) score and the American Society of Anesthesiologists (ASA) score are essential tools for the assessment of patients with various malignancies. However, doubts have arisen regarding their prognostic utility due to conflicting findings in limited studies. This study aims to comprehensively evaluate the prognostic value of preoperative ECOG-PS scores and ASA scores in patients undergoing radical nephroureterectomy (RNU) for upper tract urothelial carcinoma.

Materials and Methods:

This multicentered cohort study enrolled patients who underwent RNU with curative intentat sixteen institutes in Taiwan from 1988 to 2023. Univariable and multivariable regression analyses were used to determine the impact of ECOG-PS scores and ASA scores on survival outcomes and postoperative complications. Patients were categorized based on ECOG-PS scores (0-1 vs. 2-4) and ASA scores (1-2 vs.3-4) according to prior literature.

ELIGIBILITY:
Inclusion Criteria:

* All patients received UTUC surgery and follow-up in sixteen institutions across Taiwan

Exclusion Criteria:

* Treatment not aimed at curative intent
* Incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with UTUC and underwent RNU between 1988 and 2023, and a total of 2515 eligible patients were included in the final analysis.
Sampling Method: Non-Probability Sample
Enrollment: 2515 (Actual)
Dates: Start 1988-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1988 to 2023
  in days
Cancer-specific survival | 1988 to 2023
  in days
Disease-free survival | 1988 to 2023
  in days
Bladder recurrence-free survival | 1988 to 2023
  in days

SECONDARY OUTCOMES:
Number of patients with major postoperative complication | 1988 to 2023
  Clavien-Dindo classification grade higher or equal to III
Number of patients with postoperative renal failure | 1988 to 2023
  Those who requiring renal replacement therapy permanently

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Chih Yeh, MD, PhD, Principal Investigator — Department of Urology, Kaohsiung Medical University, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided